CLINICAL TRIAL: NCT01517750
Title: Study to Predict the Need for Humidification Use and Comparison of the Effect of ThermoSmart™ and no Humidification on Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Collaborators: Helios Klinik Ambrock (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FPH-OSA-TS-2012
Record Dates: First submitted 2012-01-18; First posted 2012-01-25 (Estimated); Results first posted 2015-06-24 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Obstructive Sleep Apnea; Humidification; Continuous Positive Airway Pressure; ICON; ThermoSmart
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- APAP with humidification (Experimental): ICON Auto CPAP™ with Thermosmart heated tube
  Interventions: Device: ICON Auto CPAP™ with Thermosmart heated tube
- APAP without humidification (Active Comparator): ICON Auto CPAP™ without Thermosmart heated tube
  Interventions: Device: ICON Auto CPAP™ without Thermosmart heated tube

INTERVENTIONS:
Device: ICON Auto CPAP™ with Thermosmart heated tube — ICON Auto CPAP™ with heated humidification and the use of a heated tube
  Arms: APAP with humidification
Device: ICON Auto CPAP™ without Thermosmart heated tube — ICON Auto CPAP™ without heated humidification or the use of a heated tube.
  Arms: APAP without humidification

SUMMARY:
Despite the effectiveness of continuous positive airway pressure (CPAP) in abolishing upper airway obstruction, acceptance of and adherence with therapy has been sub-optimal. One of the only technological advancements shown to increase adherence is heated humidification, now considered part of conventional CPAP therapy in some countries. ThermoSmart™ is a unique technology developed by Fisher & Paykel Healthcare which utilises a heated breathing tube to deliver optimal humidity in all environments. ThermoSmart has been shown to be superior to conventional humidification in reducing side effects, condensation and titrated pressure as well as increasing total sleep time. However, improved humidity delivery has not lead to significantly increased adherence in unselected obstructive sleep apnea (OSA) patients.

A total of 80 patients diagnosed with OSA but naive to CPAP use will be randomized into a single blind, randomized, parallel-arm trial to determine whether the the use of heated humidification will impact therapy adherence.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with OSA
* Naïve to CPAP therapy, i.e have not been prescribed, or used CPAP in the last 5 years
* Prescribed a nasal mask (as patients will be prescribed their mask following recruitment into the study, any participants who are prescribed a full face mask will be withdrawn)

Exclusion Criteria:

* Severe heart disease
* Co-existing lung disease
* Co-existing sleep disorders
* Pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Georg Nilius, Dr., Principal Investigator — Helios Klinik Ambrock
Locations (1):
- Helios - Klinik Ambrock, Hagen, Weg, Germany

REFERENCES:
- [Derived] Nilius G, Franke KJ, Domanski U, Schroeder M, Ruhle KH. Effect of APAP and heated humidification with a heated breathing tube on adherence, quality of life, and nasopharyngeal complaints. Sleep Breath. 2016 Mar;20(1):43-9. doi: 10.1007/s11325-015-1182-2. Epub 2015 May 10. PMID 25957615
- See also: Sponsor Site — http://www.fphcare.co.nz/

RESULTS

PARTICIPANT FLOW:
Groups:
- APAP Without Humidification + Low RIsks of NPC: ICON Auto CPAP™ (continuous positive airway pressure) without Thermosmart heated tube with patients who are classified to have a low risks (minor complaints classified as a NPC score equal or less than 9) of nasopharyngeal problems.
- APAP With Humidification + Low Risks of NPC: ICON Auto CPAP™ (continuous positive airway pressure) with Thermosmart heated tube with patients who are classified to have a low risks (minor complaints classified as a NPC score equal or less than 9) of nasopharyngeal problems.
- APAP With Humidification + High Risks of NPC: ICON Auto CPAP™ (continuous positive airway pressure) with Thermosmart heated tube with patients who are classified to have a high risks (major complaints classified as a NPC score more than 9) of nasopharyngeal problems.
- APAP Without Humidification + High RIsks of NPC: ICON Auto CPAP™ (continuous positive airway pressure) without Thermosmart heated tube with patients who are classified to have a high risks (major complaints classified as a NPC score more than 9) of nasopharyngeal problems.
Period: Overall Study
Arm/Group | APAP Without Humidification + Low RIsks of NPC | APAP With Humidification + Low Risks of NPC | APAP With Humidification + High Risks of NPC | APAP Without Humidification + High RIsks of NPC
Started | 21 | 19 | 21 | 19
Completed | 20 | 17 | 17 | 18
Not Completed | 1 | 2 | 4 | 1
Not completed — Lost to Follow-up | 1 | 2 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- APAP With Humidification + Low Risks of NPC: ICON Auto CPAP™ with Thermosmart heated tube with patients who are classified to have a low risks (minor complaints) of nasopharyngeal problems.
- APAP Without Humidification + Low RIsks of NPC: ICON Auto CPAP™ without Thermosmart heated tube with patients who are classified to have a low risks (minor complaints) of nasopharyngeal problems.
- APAP With Humidification + High Risks of NPC: ICON Auto CPAP™ with Thermosmart heated tube with patients who are classified to have a high risks (major complaints) of nasopharyngeal problems.
- APAP Without Humidification + High Risks of NPC: ICON Auto CPAP™ without Thermosmart heated tube with patients who are classified to have a high risks (major complaints) of nasopharyngeal problems.
- Total: Total of all reporting groups
Arm/Group | APAP With Humidification + Low Risks of NPC | APAP Without Humidification + Low RIsks of NPC | APAP With Humidification + High Risks of NPC | APAP Without Humidification + High Risks of NPC | Total
Number analyzed (Participants) | 17 | 20 | 17 | 18 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (9.8) | 54.3 (8.8) | 50.9 (6.8) | 52.1 (8.7) | 52.3 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 4 | 4 | 15
  Male | 15 | 15 | 13 | 14 | 57
Region of Enrollment [Number; unit: participants]
  Germany | 17 | 20 | 17 | 18 | 72

OUTCOME MEASURES:

1. Primary Outcome: Therapy Adherence With Treatment Per Night Averaged Over Total Time Period Measured Via Internal Software on the Device and Reported on Using InfoSmart™ Software With and Without Heated Humidification.
Time Frame: 6 weeks after patient randomization
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | APAP With Humidification + Low Risks of NPC | APAP Without Humidification + Low RIsks of NPC | APAP With Humidification + High Risks of NPC | APAP Without Humidification + High RIsks of NPC
Number analyzed (Participants) | 17 | 20 | 17 | 18
minutes | 330 (116) | 321 (89) | 330 (103) | 281 (118)

2. Secondary Outcome: Epworth Sleepiness Score (ESS)
Description: The ESS is a measure of daytime sleepiness and has a total of 24 points. A range from 0-9 is considered normal. A score of more than 9 is considered to have abnormal daytime sleepiness
Time Frame: 6 weeks after patient randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | APAP With Humidification + Low Risks of NPC | APAP Without Humidification + Low RIsks of NPC | APAP With Humidification + High Risks of NPC | APAP Without Humidification + High RIsks of NPC
Number analyzed (Participants) | 17 | 20 | 17 | 18
units on a scale | 5.7 (5.0) | 4.9 (4.9) | 5.7 (3.5) | 9.1 (3.9)

3. Secondary Outcome: Functional Outcome of Sleep Questionnaire (FOSQ)
Description: FOSQ is a measure of the impact of the disorder on multiple activities with everyday living and how the treatment can improve these activities. There are 30 questions and for each questions you have to pick from a subscale from 0-4; 0 = "I don't do this activity for other reasons", 1="Yes extremely", 2="Yes moderately", 3= "Yes a little", 4 = "No". Scores of each subscale will be summed up and scaled to a maximum achievable value of 20. The sum score was calculated. The value range is 0-100. A higher score means that the treatment has positively improved everyday activities.
Time Frame: 6 weeks after patient randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | APAP With Humidification + Low Risks of NPC | APAP Without Humidification + Low RIsks of NPC | APAP With Humidification + High Risks of NPC | APAP Without Humidification + High RIsks of NPC
Number analyzed (Participants) | 17 | 20 | 17 | 18
units on a scale | 91.7 (7.6) | 91.7 (14.8) | 90.0 (11.9) | 82.0 (12)

4. Secondary Outcome: Nasopharyngeal Complaints
Description: Nasopharyngeal complaints (NPC) were assessed by a questionnaire. Subjects were asked to evaluate their condition on a scale from 0 ("no complaints") to 5 ("very strong"). The following questions were asked within the questionnaire: Did you observe nasal congestion, nasal dryness, runny nose, dry mouth, and dry throat (0-5 each) during the last week. The maximal achievable sum score was 25.
Time Frame: 6 weeks after patient randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | APAP With Humidification + Low Risks of NPC | APAP Without Humidification + Low RIsks of NPC | APAP With Humidification + High Risks of NPC | APAP Without Humidification + High RIsks of NPC
Number analyzed (Participants) | 17 | 20 | 17 | 18
units on a scale | 4.4 (4.4) | 7.3 (3.1) | 5.4 (3.0) | 10.7 (6.6)

5. Post Hoc Outcome: Outcomes in Patients With ENT (Ears, Nose and Throat) Surgeries
Time Frame: 6 weeks after randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Previous ENT Surgeries + Humidification | Previous ENT Surgeries + Without Humidification | Without Previous ENT Surgeries + Humidification | WIthout Previous ENT Surgeries + WIthout Humidification
Number analyzed (Participants) | 13 | 18 | 21 | 20
units on a scale
  NPC (Nasopharyngeal complaints) | 5.0 (4.7) | 10.8 (6.1) | 4.9 (3.0) | 7.5 (4.2)
  ESS (Epworth sleepiness score) | 5.3 (5.7) | 8.1 (4.9) | 5.5 (3.2) | 6.5 (4.7)
  FOSQ (Functional outcome of sleep questionnaire | 90.9 (15.9) | 85.5 (12.1) | 90.9 (11.5) | 88.5 (10.1)

6. Post Hoc Outcome: Adherence With ENT Surgeries
Time Frame: 6 weeks after randomization
Measure: Mean (Standard Deviation); unit: mins
Arm/Group | Previous ENT Surgeries + Humidification | Previous ENT Surgeries + Without Humidification | Without Previous ENT Surgeries + Humidification | WIthout Previous ENT Surgeries + WIthout Humidification
Number analyzed (Participants) | 13 | 18 | 21 | 20
mins | 327.9 (121.1) | 285.6 (124.6) | 331.5 (102.2) | 317.0 (82.8)

ADVERSE EVENTS:
Arm/Group | APAP With Humidification + Low Risks of NPC | APAP Without Humidification + Low RIsks of NPC | APAP With Humidification + High Risks of NPC | APAP Without Humidification + High RIsks of NPC
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21 | 1/21 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/21 | 0/21 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APAP With Humidification + Low Risks of NPC (N=19) | APAP Without Humidification + Low RIsks of NPC (N=21) | APAP With Humidification + High Risks of NPC (N=21) | APAP Without Humidification + High RIsks of NPC (N=19)
Hospitalization for Ureter Obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated event that was resolved with no sequel at the end of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No